CLINICAL TRIAL: NCT06837220
Title: Enhancing the Implementation of Tobacco Treatment: A Community-responsive Approach
Brief Title: Implementation of Tobacco Cessation Programming at Community Behavioral Health Sites
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Respiratory Health Association (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-2154; P50MD017349 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Nicotine Use Disorder; Smoking Cessation; Smoking Cessation Intervention
Keywords: smoking; smoking cessation; nicotine; nicotine use disorder; quitting smoking; quitting nicotine; respiratory health; telehealth; virtual; tobacco; tobacco treatment; community; behavioral health; chicago; group therapy; disparities; adults who smoke; cigarettes; tobacco cessation; cessation; abstinence; substance use; substance abuse; addiction; counseling; health counseling; health communication
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking; Tobacco Use Cessation; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Intervention (Experimental): The participants in this arm will take part in a pilot test of a community-targeted smoking cessation treatment. This treatment will be evidence-based smoking treatment using cognitive behavioral and motivational strategies implemented according to findings from Phase 1 of this study. The original intervention has four core sessions that will be modified accordingly to fit community needs. Participants will complete pre- and post-session questionnaires regarding their smoking status, quit attempts, use of smoking cessation aids, and other surveys.
  Interventions: Behavioral: Enhanced Courage to Quit

INTERVENTIONS:
Behavioral: Enhanced Courage to Quit — Participants will engage in a version of the smoking cessation treatment "Courage to Quit" that has been optimized for implementation in community behavioral health clinics. The group will run over a period of 3 months, where participants will learn behavioral and cognitive skills for smoking cessation and/or reduction. Special attention will be given to the unique needs of the community, such as technology options or more flexible treatment models. The goal of this intervention is to prove that it is feasible to implement, and can create enhanced engagement and smoking outcomes for adults who smoke (AWS) and have fewer socioeconomic resources.

SUMMARY:
The goal of this study is to: partner with Respiratory Health Association and determine barriers and unmet smoking cessation treatment needs from leaders in behavioral health organizations, treatment programs and adults who smoke (AWS) in Chicago. This will be accomplished by establishing a community advisory board (CAB) and pilot testing a community-informed smoking cessation treatment within a community behavioral health organization to determine its feasibility after addressing implementation issues.

DETAILED DESCRIPTION:
The purpose of the proposed study is to determine barriers and unmet smoking cessation treatment needs from leaders in behavioral health organizations, behavioral health treatment providers, and community members in Chicago and pilot test a community-informed, targeted rolling smoking cessation treatment within a community organization. The research team and the Respiratory Health Association (RHA) will work together to identify community sites that could derive possible benefit from adopting and implementing the targeted treatment.

Aim 1: Develop a Community Advisory Board (CAB) comprised of providers, community members, and organization leadership.

Aim 2: Use a mixed-methods approach to understand barriers, facilitators, and unmet treatment needs regarding smoking cessation treatment within the community.

Aim 3: Pilot test the targeted smoking cessation treatment across a 3-month period at one community site through partnership with Respiratory Health Association.

Hypothesis: The targeted intervention will demonstrate feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Identify as someone who currently smokes combustible cigarettes (at least 1 cigarette per day) on each day for the past month
* Report interest in quitting cigarettes (at least 6/10 scale in interest of quitting)
* Age 18 or older, ability to understand the English language, willing and able to provide informed consent
* Stable residence and contact information throughout the follow up period

Exclusion Criteria:

* Non-daily or intermittent cigarette use
* No interest in quitting smoking
* Unstable residence/not staying in Chicago for duration of study period
* Current untreated severe substance use disorder (with the exception of tobacco use) or past-year serious untreated psychiatric illness (e.g. schizophrenia, bipolar disorder, obsessive compulsive disorder, unspecified psychosis, past-year suicide attempt)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who attend the enhanced intervention as assessed by enrollment and sign-in at each session | 3 months
  Investigators will consider the initial pilot period of the enhanced intervention successful if the team enrolls (attend one session) and retains (attend four or more sessions) at least three participants in the pilot treatment across three months
Feasibility will be assessed by calculating the portion of people who enroll (attend at least on session) and complete 4+ sessions versus those who drop out before finishing 4 sessions as assessed by session sign-in | 3 months
  Investigators will consider the intervention design to be feasible if fewer than 40% of enrollees drop out after their first attended session.
A modified version of the Client Satisfaction Questionnaire (CSQ) will assess intervention acceptability. | End of treatment (e.g., 3 months or fourth session attended, whichever comes first)
  This measure is a 10-point Likert scale (0=not at all, 10=very much) that assesses items such as intervention quality, effectiveness, and intrusiveness. For acceptability, the study team predicts at least 75% of participants will rate the intervention as acceptable via post-treatment survey (CSQ).

SECONDARY OUTCOMES:
Change in number of cigarettes consumed per day | Through study completion, an average of 3 months
  Participant self-report of past week average cigarettes smoked per day
Use of nicotine replacement therapy and FDA-approved cessation medication | Through study completion, an average of 3 months
  Participant self-report of pharmacotherapy will be assessed at each session and end of treatment
Number of quit attempts | Through study completion, an average of 3 months
  The number of times each participant has tried to quit, whether successful or not
Motivation to change smoking behavior via Contemplation Ladder | Through study completion, an average of 3 months
  Participants' interest in quitting will be assessed on a 10-point quit interest scale (e.g., The Contemplation Ladder). Scores range from 0-10 with higher scores indicating greater motivation to change.

IPD SHARING:
Plan to Share IPD: Undecided